CLINICAL TRIAL: NCT05765175
Title: Cardiac RADIoablation Versus Repeat Catheter Ablation: a Pivotal Randomized Clinical Trial Evaluating Safety and Efficacy for Patients With High-risk Refractory Ventricular Tachycardia
Brief Title: Cardiac RADIoablation Versus Repeat Catheter Ablation: a Pivotal Randomized Clinical Trial Evaluating Safety and Efficacy for Patients With High-risk Refractory Ventricular Tachycardia (RADIATE-VT)
Acronym: RADIATE-VT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAR-2022-01
Record Dates: First submitted 2023-02-15; First posted 2023-03-13 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Tachycardia, Ventricular
Keywords: Cardiac radioablation; Ventricular tachycardia; Catheter ablation; Refractory ventricular tachycardia; High risk; SBRT
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: The Varian CRA trial is a multicenter, international, pivotal, 2-arm randomized controlled trial (RCT). Subjects will be randomized 1:1 to CRA or repeat CA. Randomization will be stratified by (1) enrolling institution and (2) NYHA class I/II vs. III/IV. Blinding will not be used in this trial, as the different interventions cannot be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Repeat catheter ablation (CA) (Active Comparator)
  Interventions: Procedure: Catheter Ablation (CA)
- Varian Cardiac Radioablation (CRA) (Experimental)
  Interventions: Device: Varian Cardiac Radioablation (CRA)

INTERVENTIONS:
Device: Varian Cardiac Radioablation (CRA) — Subjects randomized to CRA will be treated with the Varian CRA system according to a uniform CRA protocol. A dose of 25 Gy in a single fraction is prescribed to the planning target volume (PTV), and delivered using a stereotactic body radiotherapy (SBRT) technique.
  Arms: Varian Cardiac Radioablation (CRA)
Procedure: Catheter Ablation (CA) — Subjects randomized to the CA arm will be treated according to a uniform CA protocol.
  Arms: Repeat catheter ablation (CA)

SUMMARY:
RADIATE-VT is a pivotal, multicenter, randomized trial comparing safety and efficacy between cardiac radioablation (CRA) using the Varian CRA System and repeat catheter ablation (CA), for patients with high-risk refractory ventricular tachycardia (VT) who have experienced VT recurrence after CA and are candidates for additional CA.

ELIGIBILITY:
Inclusion Criteria:

1. High-risk refractory VT, defined as:

   1. Ischemic and/or nonischemic cardiomyopathy, and
   2. Recurrent sustained monomorphic VT, defined as at least one of the following below, documented by ICD interrogation or ECG in the prior 6 months, and having occurred after the last VT ablation:

      A: ≥3 episodes of monomorphic VT treated with anti-tachycardia pacing (ATP) at least one of which is symptomatic

      B: ≥1 appropriate ICD shock

      C: ≥3 episodes of sustained monomorphic VT within 24 hours treated with ICD shock or ATP

      D: sustained monomorphic VT below detection rate of ICD documented by ECG, and
   3. Left ventricular ejection fraction (LVEF) ≤49% and
   4. Previously underwent at least one standard of care CA for VT.
2. Presence of a clinical indication for a repeat CA procedure for scar-mediated VT in the judgement of the treating investigator.
3. Has failed amiodarone therapy or is intolerant to amiodarone:

   * Failed amiodarone therapy is defined as: appropriate ICD therapy or sustained monomorphic VT having occurred while the patient was taking amiodarone (minimum cumulative dose of 10 g).
   * Intolerant to amiodarone is defined as: previously tried or taken amiodarone but stopped due to medication related side effects or toxicities.
4. Deemed to be medically and technically a candidate for further CA by the electrophysiologist investigator.
5. Presence of an ICD.
6. At least 18 years of age (or meets local age of majority).
7. Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

1. Contraindication to a CA procedure for VT (e.g., presence of mobile LV thrombus, active systemic infection, active ischemic or other reversible causes of VT).
2. Patients with expected, right ventricular scar only.
3. Any prior radiation to the thorax region of the body.
4. Known medical conditions associated with higher risk of radiotherapy complications in the judgement of the radiation oncologist (i.e., active connective tissue disorders, interstitial lung disease, etc.) that would preclude safe delivery of CRA.
5. Current use of inotropes.
6. Presence of a left-ventricular assist device (LVAD).
7. Scheduled for LVAD or heart transplant procedures.
8. Presence of a systemic illness likely to limit survival to < 1 year.
9. VT ablation procedure performed within the prior 2 weeks.
10. Polymorphic VT or ventricular fibrillation (VF) as the primary clinical heart rhythm, as indicated by 12-lead ECG and/or ICD interrogation.
11. >3 distinct clinical monomorphic VT morphologies on ICD interrogation since the prior CA, or >5 induced monomorphic VT morphologies during NIPS testing.
12. Incessant VT that is hemodynamically unstable.
13. Bundle branch reentry (BBR) VT.
14. Pregnant and/or breastfeeding. (Patient denial is sufficient for enrollment).
15. Patients of childbearing potential who:

    * are not on a medically effective means of birth control at the time of screening or do not start a medically effective means of birth control prior to randomization; or
    * do not agree to continue medically effective means of birth control until they have completed their assigned therapy; or
    * do not agree to be on a medically effective means of birth control if they are treated with CRA after their index CA procedure.
16. Patients enrolled in another clinical study the investigator believes to be in conflict with this clinical investigation.
17. Patients enrolled or planned to be enrolled in another cardiac radioablation clinical study or registry.
18. Patients with any other medical condition or laboratory value that would, at the discretion of the investigator, preclude the patient from participation in this clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Co-primary safety endpoint: freedom from treatment-attributed (i.e., probably or definitely related) serious adverse events (SAEs) | Treatment through 12 months post-treatment
  Freedom from treatment-attributed (i.e., probably or definitely related) serious adverse events (SAEs), evaluated from treatment through 12 months post-treatment.
Co-primary efficacy endpoint: Freedom from death, and appropriate ICD shock, and VT storm. | Death will be counted from randomization through 12 months, and shock and storm will be counted starting after a 30-day period immediately post-randomization and continuing through 12 months post randomization
  Freedom from death, and appropriate ICD shock, and VT storm, where death will be counted from randomization through 12 months, and shock and storm will be counted starting after a 30-day period immediately post-randomization and continuing through 12 months post randomization.

SECONDARY OUTCOMES:
Change in quality of life at 6 weeks post treatment: | From baseline through 6 weeks post treatment
  Change in quality of life at 6 weeks post treatment measured by the Short Form Health Survey 36 (SF-36) Health Change Question. This item asks the subject to rate their health in general compared to one year ago in a 5-point scale of 1 (much better), 2 (somewhat better), 3 (about the same), 4 (somewhat worse), 5 (much worse).
VT burden reduction | From 6 months before randomization through to a 6 month period starting after a 30-day period immediately post-randomization
  VT burden reduction measured as a ≥75% reduction in appropriate ICD therapies (ATP, shock), comparing a 6-month period before randomization and a 6-month period starting after a 30-day period immediately post-randomization.
Change in quality of life (Social Functioning) at 6 weeks post treatment | From baseline through 6 weeks post treatment
  Change in quality of life (Social Functioning) measured by the Short Form Health Survey 36 (SF-36) Social Functioning item (social activities in past 4 weeks). This item asks the subject to rate how much of the time their physical health or emotional problems interfered with their social activities in the past 4 weeks in a 5-point scale of 1 (All of the time), 2 (Most of the time), 3 (Some of the time), 4 (A little bit of the time), 5 (None of the time).

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Hartford Hospital, Hartford, Connecticut
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - The Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No